CLINICAL TRIAL: NCT02225873
Title: The Effectiveness of Two Training Protocols When Managing Chronic Cervical Pain: Controlled Randomized Clinical Trial.
Brief Title: The Effectiveness of Exercises Protocol in Management of Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Dr., University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2013/046/20140528
Record Dates: First submitted 2014-08-24; First posted 2014-08-26 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Proprioception

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- strength-endurance exercises (Experimental): Group 1 (experimental) will carry out motor control exercises through cranio-cervical flexion training and strength-endurance exercises.
  Interventions: Other: motor control exercises
- strength-endurance and proprioception (Placebo Comparator): Group 2 (control) will carry out exercises to improve muscle strength-endurance and proprioception.
  Interventions: Other: muscle strength-endurance and proprioception

INTERVENTIONS:
Other: motor control exercises — Will carry out intermuscular coordination exercises through cranio-cervical training, following Jull et al. and exercises to increase strength-endurance on the neck flexor muscles
  Arms: strength-endurance exercises
Other: muscle strength-endurance and proprioception — Will carry out proprioception exercises through articular repositioning training and exercises to increase strength-endurance on the neck flexor muscles. They will be performed in the same way as the experimental group protocol.
  Arms: strength-endurance and proprioception

SUMMARY:
This study will verify whether the cranio-cervical flexion coordination (motor control) and muscle strength training protocol is more effective in improving muscle than the proprioception and muscle strength protocol in patients with chronic neck pain.

Hypothesis: The craniocervical flexion (motor control) and muscle strength training protocol will improve muscle function more than the proprioception and muscle strength protocol in patients with chronic cervical pain.

Objective: To find out if applying the strength therapeutic exercise protocol and the craniocervical flexion coordination (motor control) training is more effective than the strength and articular repositioning protocol when carrying out the craniocervical flexion test in patients with chronic cervical pain.

DETAILED DESCRIPTION:
Neck pain is delimited by two horizontal lines, one through the lower portion of the occipital region and one through the spinous process of the first thoracic vertebra. This pain is reproduced by neck movements or exploratory provocation tests. Scientific studies show that at least two out of three people will experience neck pain throughout life. Some of the causes are traumatism and whiplash although sometimes pain is idiopathic.

This study will verify whether the cranio-cervical flexion coordination (motor control) and muscle strength training protocol is more effective in improving muscle than the proprioception and muscle strength protocol in patients with chronic neck pain.

The project design will be a randomized controlled evaluator-blinded clinical trial with two intervention groups:

Group 1 (experimental) will carry out motor control exercises through cranio-cervical flexion training and strength-endurance exercises.

Group 2 (control) will carry out exercises to improve muscle strength-endurance and proprioception. Measurements will be done at the beginning of the study, pre and post-treatment, one month and two months after treatment and throughout the six month treatment. Each session will last 45 minutes and therapy will be performed without provoking the patient symptoms.

Intervention

Experimental group 1: will carry out intermuscular coordination exercises through cranio-cervical training, following Jull et al1, 2 and exercises to increase strength-endurance on the neck flexor muscles.

Control group 2: will carry out proprioception exercises through articular repositioning training and exercises to increase strength-endurance on the neck flexor muscles. They will be performed in the same way as the experimental group protocol.

ELIGIBILITY:
Inclusion Criteria:

* History of cervical pain of at least 3 months.
* Between 18 and 55 years old.
* Altered movement and/or loss of cervical control.
* Pain after palpation of the muscles to be treated.

Exclusion Criteria:

* Previous history of central neurological condition.
* Previous surgery of the cervical, cranial, scapular waist, upper limb or jaw.
* Having received specific treatment or therapy of the cervical region in the 6 months prior to the study.
* Neck pain or headache with no musculo-skeletal causes.
* Any other disorder that prevents physical activity.
* Having received psychological treatment due to neck pain.
* Patients with fibromyalgia, rheumatoid arthritis, vascular diseases, neoplasm or vestibular system pathologies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Craniocervical Flexion Test | up to six months after treatment
  This test measures the activation and resistance of the neck flexor muscles in 5 steps, with isometric contractions on the patient every 2 mmHg, increasing pressure sequentially from 20 mmHg up to 30 mmHg.
  Once carried out the test, performance will be measured by the pressure level achieved and the number of times pressure can be maintained by the patient with the correct cranioflexion movement in each level.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Gallego-Izquierdo, Dr, Study Chair — Alcala University
Locations (1):
- Alcalá University, Alcalá de Henares, Madrid, Spain